CLINICAL TRIAL: NCT02923973
Title: Transvaginal Ultrasound Cervical Length Screening in Singleton Pregnancy With Prior Spontaneous Preterm Birth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Pisa - Prof Paolo Mannella (Unknown)
Responsible Party: Principal Investigator, Gabriele Saccone, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #30/18
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVU CL screening (Experimental): TVU CL screening: serial TVU CL scan from 16 0/7 to 24 6/7 every week, for a total of nine scans Vaginal progesterone 200mg suppository daily from 14 0/7 to 20 6/7 weeks for the history of prior spontaneous preterm delivery
  Interventions: Other: Transvaginal ultrasound cervical length screening
- No TVU CL screening (No Intervention): no screening Vaginal progesterone 200mg suppository daily from 14 0/7 to 20 6/7 weeks for the history of prior spontaneous preterm delivery

INTERVENTIONS:
Other: Transvaginal ultrasound cervical length screening — Serial transvaginal ultrasound cervical length scan every week from 16 to 24 weeks
  Arms: TVU CL screening

SUMMARY:
Preterm birth (PTB) is the major cause of perinatal morbidity and mortality. Worldwide, about 15 million babies are born too soon every year, causing 1.1 million deaths, as well as short- and long-term disability in countless survivors. Few prognostic tests are available to predict PTB. A short transvaginal ultrasound cervical length (TVU CL) has been shown to be a good predictor of PTB.Different strategies have been adopted for prevention of PTB. The evidence supports the use of vaginal progesterone in singleton pregnancies with short cervix, while cervical cerclage seems to be beneficial only in the subgroup of singleton gestations with both prior spontaneous PTB and TVU CL ≤25mm, and not in singletons without prior PTB, nor in multiple gestations.

However, so far there are no level-1 data on the efficacy of TVU CL screening neither in low risk nor in high risk pregnancy Thus, the investigators aim to assess the efficacy of a policy of TVU CL screening in singleton pregnancy with prior spontaneous PTB

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Singleton gestations
* Women with prior spontaneous preterm birth, defined as spontaneous preterm delivery 16 0/7 - 36 6/7 weeks

Exclusion Criteria:

* multiple gestation
* Ruptured membranes or fetal structural or chromosomal abnormality at the time of randomization
* Ballooning of membranes outside the cervix into the vagina at the time of randomization
* Labor or cerclage in situ at the time of randomization

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Less than 37 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
preterm birth rates | Less than 24, 28, 34 weeks gestation
Birth weight | Time of delivery
Low birth weight | Time of delivery
  Birth weight <2500g
Neonatal death | Between birth and 28 days of age
Composite adverse neonatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis and neonatal death
Admission to neonatal intensive care unit | Between birth and 28 days of age

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gabriele Saccone, Naples
  - University of Pisa, Pisa